CLINICAL TRIAL: NCT01951430
Title: Observational Prospective Multicenter Study to Evaluate the Infective Risk in Myelodysplastic Syndrome Patients: Antimicrobial Prophylaxis and Granulocyte Growth Factors.
Brief Title: Observational Evaluation of Infective Risk in Myelodysplastic Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: MDS0413
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: Adult patients; Infective events; Antibiotic; Antifungal; Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Anti-Bacterial Agents; Antifungal Agents; Ofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Cephalosporins; posaconazole; Fluconazole; Itraconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myelodysplastic syndrome patients: Patients affected by myelodysplastic syndrome enrolled in the observational study
  Interventions: Drug: Antibiotic and antifungal drugs

INTERVENTIONS:
Drug: Antibiotic and antifungal drugs
  Other Names: levofloxacine;; cyprofloxacine;; co-trimoxazole;; chinolones;; cephalosporins;; penicillines;; other betalactams;; macrolids;; posaconazole;; fluconazole;; itraconazole.

SUMMARY:
The purpose of this study is to observe the number of new cases of infections per population in a given time period and their characteristics in a pathology (myelodysplastic syndrome, MDS)that involves ineffective production (or dysplasia) of a class of blood cells.

DETAILED DESCRIPTION:
The scarcity and the inadequacy of data make impossible the writing of evidence-based recommendations for prevention and management of infections in myelodysplastic syndrome.

The aim of this study is to evaluate the incidence and the spectrum of the infections of MDS patients. Will be also evaluated potential risk factors.

This study could help the definition of the optimal management of MDS patients in terms of prophylaxis of the infective complications and in terms of the correct administration of growth factors.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years) with newly diagnosed myelodysplastic syndrome or patients who have undergone a bone marrow reevaluation;
* Signed written informed consent;

Exclusion Criteria:

* Psychiatric patients;
* Patients with life expectancy less than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult myelodysplastic syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2014-03; Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Number of infectious events in myelodysplastic syndrome patients | at 1 year from study entry
  Infectious events are fungal and antibiotic events

SECONDARY OUTCOMES:
Number of MDS patients with a febrile event treated with antibiotic, antifungal and antiviral therapy | at 1 year from study entry
Level of neutropenia | at 1 year from study entry
Number of patients who recover from infection | at 1 year from study entry
Number of patients recovered from infection out of the total of patients with documented infection during the observational period | at 1 year from study entry
Number of patients who don't develop bacterial infection | at 1 year from study entry
Number of patient who don't develop fungal infection | at 1 year from study entry
Number of patient who don't develop viral infection | at 1 year from study entry
Number of patients that needed granulocyte growth factors | at 1 year from study entry
Number of patients that needed iron sequestrating therapy caused by iron overload | at 1 year from study entry
Length of the hospitalization | at 1 year from study entry
Weeks of MDS suspension treatment | at 1 year from study entry
Number of patients responding to therapy according to the administered treatment | at 1 year from study entry
Number of MDS patients alive | at 1 year from study entry
Number of patients without MDS progression | at 1 year from study entry
Need for hospitalization | at 1 year from study entry
Level transfusion dependence | At one year from study entry
Level of MDS subtype | At one year from study entry
Level of risk of International Prognostic Scoring System (IPSS) | At one year from study entry
Level of International Prognostic Scoring System (IPSS)-revised | At one year from study entry
Level of iron overload | At one year from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Livio Pagano, Dr., Principal Investigator — Università Cattolica del Sacro Cuore - Policlinico A. Gemelli - Roma
Locations (25):
- Italy (25):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale 'Torrette', Ancona
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Divisione di Ematologia Ospedale A. Perrin, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Policlinico di Careggi, Florence
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Med. Int. ed Oncologia Medica IRCCS Policlinico S. Matteo, Pavia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari Azienda Ospedaliero-Universitaria, Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.gimema.it